CLINICAL TRIAL: NCT01156259
Title: Phase 3 Study of 30Gy Versus 40Gy Involved-field Radiotherapy in Localized Diffuse Large B Cell Lymphoma Achieving CR After Chemotherapy
Brief Title: 30Gy Versus 40Gy Involved-field Radiotherapy for Localized Diffuse Large B Cell Lymphoma Achieving CR After Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Department of Radiation Oncology, Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-LYM-004
Record Dates: First submitted 2010-06-29; First posted 2010-07-02 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-04

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: B cell cll/lymphoma, human
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 30 Gy (Experimental)
  Interventions: Radiation: 3D-CRT based Involved Field Radiotherapy
- 40 Gy (Active Comparator)
  Interventions: Radiation: 3D-CRT based Involved Field Radiotherapy

INTERVENTIONS:
Radiation: 3D-CRT based Involved Field Radiotherapy — CT simulation, 3D-CRT or IMRT techniques, Involved Field Radiotherapy of 30Gy
  Arms: 30 Gy
Radiation: 3D-CRT based Involved Field Radiotherapy — CT simulation, 3D-CRT or IMRT techniques, Involved Field Radiotherapy of 40Gy
  Arms: 40 Gy

SUMMARY:
The purpose of this study is to determine whether 30Gy Involved-field Radiotherapy (IFRT) is as effective as 40Gy in the treatment of localized Diffused Large B cell Lymphoma (DLBCL) when completing CR after chemotherapy.

DETAILED DESCRIPTION:
The best proper doses of IFRT in combined modality treatments (CMT) for localized DLBCL is still undetermined. Existing treatment guidelines recommend 40Gy or above as the standard treatment dosage. However, there were large-scaled clinical trials implying smaller doses such as 30Gy may be equivalent effective. Lowering radiation doses can decrease treatment toxicities and radiotherapy-induced diseases, which has been conformed by HD13 study for Hodgkin's Lymphoma. It may even retain the truth when modern era radiation techniques are involved and especially in patients achieving CR after chemotherapy. A comprehensive, prospective dose-comparing study is needed.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-proved Diffuse Large B cell lymphoma
* nonbulky stage I, nonbulky stage IE, nonbulky stage II, or nonbulky stage IIE disease(Bulky disease was defined as a mass 10 cm or more in maximal diameter) according to Ann Arbor Staging
* provide written informed consent
* Complete regression after chemotherapy
* Considerable to CT simulation and 3D CRT or IMRT
* Performance status 0-2 WHO criteria；life expectation>6 months
* negative for human immunodeficiency virus syndrome (HIV)
* Minimal staging included chest radiograph, computed tomography of the abdomen and pelvis, and single percutaneous bone marrow biopsy and blood studies

Exclusion Criteria:

* primary mediastinal large B cell lymphoma
* dermatological lymphoma
* testicular lymphoma
* primary central nerve system lymphoma
* prior RT
* history of low-grade lymphoma congestive
* history of heart failure (CHF; New York Heart Association [NYHA] classifications III-IV), history of neoplasm (adequately treated basal cell carcinoma of the skin or in situ carcinoma of the uterine cervix were allowed), abnormal liver function tests (aminotransferases and alkaline phosphatase > 2.5 times the upper limit of normal, bilirubin > 50 ), renal insufficiency (serum creatinine > 300 ), and patients with any serious medical or psychiatric illness that would prevent informed consent or completion of protocol-prescribed treatment and follow-up

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
disease free survival | five years

SECONDARY OUTCOMES:
overall survival | five years
acute treatment toxicity | up to 16 weeks
late treatment toxicity | five years
treatment failure type | five years

CONTACTS AND LOCATIONS:
Overall Officials: Yexiong Li, MD, Study Director — Department of Radiation Oncology, Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China